CLINICAL TRIAL: NCT04363372
Title: A Pilot, Multiple Dose Study to Evaluate the Efficacy and Safety of MRx-4DP0004 in Hospitalised Patients With Symptoms of COVID-19 (SARS-CoV-2 Infection)
Brief Title: A Study for Efficacy and Safety of Live Biotherapeutic MRx4DP0004 to Treat COVID-19
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment Issues
Sponsor: 4D pharma plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MRx-4DP0004-II-001
Record Dates: First submitted 2020-04-24; First posted 2020-04-27 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2020-06

CONDITIONS: COVID-19
Keywords: MRx-4DP0004; Coronavirus; Live Biotherapeutic Product; SARS-CoV-2; Immunomodulatory
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MRx-4DP0004 (Experimental): Patients receiving standard of care will add MRx-4DP0004 to their treatment. MRx-4DP0004 is taken as 2 capsules, twice a day for 14 days. Daily dose is 4 x 10^9 to 4 x10^10 colony forming units.
  Interventions: Drug: MRx-4DP0004
- Placebo (Placebo Comparator): Patients receiving standard of care will also take 2 placebo capsules, twice a day for 14 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MRx-4DP0004 — MRx-4DP0004 is a lyophilised formulation of a proprietary strain of bacteria.
  Arms: MRx-4DP0004
Drug: Placebo — Placebo capsules will be identical in appearance to active product.
  Arms: Placebo

SUMMARY:
This is a randomised, double-blind, placebo controlled study to evaluate the efficacy and safety of MRx-4DP0004 in patients with COVID-19.

90 hospitalised patients will be enrolled and randomised (2:1) to receive MRx-4DP0004 or placebo for up to 14 days.

MRx-4DP0004 is an immunomodulating Live Biotherapeutic Product (LBP) which is expected to prevent or reduce the hyperinflammatory response to SARS-CoV-2 infection without impairing viral clearance.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to sign the consent form
* Suspected or confirmed COVID-19 as defined by:

  1. Positive RNA test for SARS-CoV-2 OR
  2. Presenting with symptoms of COVID-19 as determined by the investigator, and
  3. A score of 4 or 5 on the WHO Ordinal Scale for Clinical Improvement, and
  4. Oxygen saturation of <95% on room air, and
  5. Chest X-ray with evidence of COVID-19 e.g. ground-glass opacities
* Requires admission to hospital
* Able to swallow oral capsules

Exclusion Criteria:

* Known valvular heart defects, pulmonary hypertension or heart failure
* Known to have cystic fibrosis
* GI fistula or malabsorption syndrome
* Known allergy to ampicillin, clindamycin and imipenem
* Any other condition which, in the opinion of the investigator, would prevent full participation in the study or would interfere with the evaluation of the study endpoints
* Antibiotic treatment at enrolment or within 2 days prior
* Pregnant or breastfeeding females
* Unable or unwilling to follow contraception requirements
* Concurrent participation in another interventional clinical trial at enrolment or within 30 days prior

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-08 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Change in mean clinical status score in each treatment arm | Baseline to Day 42
  Clinical status score will be measured using the WHO Ordinal Scale for Clinical Improvement where patients are scored on a scale of 0-8 with 0 being uninfected and 8 being dead

SECONDARY OUTCOMES:
Number of adverse events in each treatment arm | Baseline to Day 42
  Safety and tolerability will be determined according to clinically relevant reported adverse events
Number of patients with an improvement in clinical status score in each treatment arm | Day 1 to Day 42
  Point changes in clinical status score will be measured using the WHO Ordinal Scale for Clinical Improvement
Number of patients with a deterioration in clinical status score in each treatment arm | Day 1 to Day 42
  Point changes in clinical status score will be measured using the WHO Ordinal Scale for Clinical Improvement
Number of patients with at least 95% oxygen saturation on room air in each treatment arm | Day 1 to Day 14
  Oxygen saturation will be measured as per local standard procedures
Time to patients with at least 95% oxygen saturation on room air in each treatment arm | Day 1 to Day 14
  Oxygen saturation will be recorded daily during hospitalisation to determine the mean time for each arm to reach at least 95% saturation
Number of patients with an improvement in the National Early Warning Score (NEWS) 2 in each treatment arm | Day 1 to Day 14
  The NEWS 2 is based on aggregate scoring of physiological measurements including respiration rate, oxygen saturation, systolic blood pressure, pulse rate, level of consciousness and temperature
Number of patients with an deterioration in the National Early Warning Score (NEWS) 2 in each treatment arm | Day 1 to Day 14
  The NEWS 2 is based on aggregate scoring of physiological measurements including respiration rate, oxygen saturation, systolic blood pressure, pulse rate, level of consciousness and temperature
Number of patients requiring Continuous Positive Airway Pressure in each treatment arm | Day 1 to Day 14
  Details of required respiratory support will be recorded throughout hospitalisation
Number of patients requiring Intermittent Positive Pressure Ventilation in each treatment arm | Day 1 to Day 14
  Details of required respiratory support will be recorded throughout the treatment period
Time to patients requiring Continuous Positive Airway Pressure in each treatment arm | Day 1 to Day 14
  Details of required respiratory support will be recorded throughout the treatment period
Time to patients requiring Intermittent Positive Pressure Ventilation in each treatment arm | Day 1 to Day 14
  Details of required respiratory support will be recorded throughout the treatment period
Time to discharge in each treatment arm | Day 1 to Day 42
  Length of hospital stay will be compared
Number of deaths in each treatment arm | Day 1 to Day 42
  All cause mortality will be compared

CONTACTS AND LOCATIONS:
Overall Officials: Dinesh Saralaya, MBBS, MD, MRCP, FRCP, Principal Investigator — Bradford Royal Infirmary
Locations (1):
- University Hospitals Plymouth NHS Trust, Plymouth, United Kingdom

IPD SHARING:
Plan to Share IPD: No